CLINICAL TRIAL: NCT05116527
Title: Pilot FMRI Studies of THC Effects on Memory and Reward Learning
Brief Title: THC Memory & Reward Learning Pilot
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, Godfrey Pearlson, Founding Director Olin Neuropsychiatry Research Center; Professor Yale University, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: HHC-2021-0195
Record Dates: First submitted 2021-10-28; First posted 2021-11-11 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-04

CONDITIONS: Marijuana; THC; Cannabis
Keywords: Cannabis; THC; Marijuana; MRI; Memory; Learning
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols; Dronabinol

STUDY DESIGN:
Intervention Model Description: All subjects will receive both study drug and placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Dose THC (Experimental): Participants will receive high dose THC.
  Interventions: Drug: Marijuana, Hash, THC, or Grass
- Placebo THC (Experimental): Participants will receive placebo THC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Marijuana, Hash, THC, or Grass — Marijuana flower with a high THC content
  Other Names: Marijuana; THC
  Arms: High Dose THC
Drug: Placebo — Placebo THC - marijuana flower with no THC content
  Arms: Placebo THC

SUMMARY:
Tetrahydrocannabidiol (THC) is the psychoactive chemical in cannabis that makes people high. This study aims to dissect acute impairment of various forms of memory and learning by THC in cannabis compared to placebo. Impairment will be assessed via a short cognitive test battery and then subjects will complete four tasks in the fMRI scanner.

DETAILED DESCRIPTION:
The protocol below is designed to begin dissecting acute impairment of various forms of memory and learning by THC in cannabis compared to placebo, in a 2-session per subject double-blind, random assignment, placebo-controlled counterbalanced design in young to middle-aged adults. The purpose of these experiments is to gather important pilot data to demonstrate proof of principle for a planned NIDA submission of a P50 center application that will examine cannabis's differential effects on the neural circuit underpinnings these various cognitive domains across the lifespan in much more detail. In other words, these pilot data will show NIDA that the investigators' methods and approaches work and are suitable for use in their proposed center grant application. Unlike in the planned P50, in these small-scale pilot studies the investigators are only concerned with comparing these disrupting effects using a single dose of THC versus placebo, without exploration of age, sleep, or sex-related differential effects or of different dose-related effects.

Tasks tapping each of the major cognitive memory-related domains will be performed in the MRI scanner, to reveal the relevant underlying circuitry and its disruption by drug using functional MRI. Although each of the fMRI tasks is already implemented in the investigators' lab in other contexts, the investigators have never studied alteration of the fMRI tasks by THC. Neither have other investigators elsewhere used this approach. It is also important to point out that the dose of active THC to be administered is the same as that already used safely in the investigators' IRB-approved driving studies, one which subjects state subjectively (a blind to actual dose information) makes them feel moderately intoxicated, and similar to the amount that they would consume themselves recreationally.

The study will consist of 3 days (screening visit and 2 dose days). In a randomized, counterbalanced, double-blind study, investigators will administer high THC marijuana or placebo marijuana using paced inhalation through a vaporizer. Following administration, subjects will provide subjectively-rated CNB intoxication using a verbal analog scale, a short cognitive test battery, then complete 4 fMRI paradigms within ~1.5 hours: a) MSDM task, b) MID task, c) RISE task, and d) Treadway Effort/Reward task. These tests will be counterbalanced across subjects and sessions to minimize order and fatigue effects.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years old
* Right handed
* CNB use within past 2 years and felt "high" when used
* Able to read, speak, and understand English
* Able and willing to provide written informed consent, and willing to commit to study protocol.

Exclusion Criteria:

* Current marijuana tolerance, desire to cut down, or cravings to sue during periods of abstinence.
* Strongly left-handed
* Positive screen for drug or alcohol (except CNB) on test day will result in rescheduling the appointment
* History of adverse effects with CNB
* CNB users who are abstaining
* Report of any psychotic disorder in a first degree relative
* IQ < 80 on the Wechsler Abbreviated Scale of Intelligence
* Inability to comprehend written instructions using the WRAT-4 reading achievement test
* Pregnant, breastfeeding, and ineffective birth control methods.
* Unable or unsafe to have an MRI
* Serious medical, neuro-ophthalmological, or neurological illness (e.g. cancer, seizure disorders, encephalopathy
* History of head trauma with loss of consciousness > 30 minutes or concussion lasting 30 days.
* Focal brain lesion seen on structural MRI
* Any medical/neurological condition that could compromise neurocognitive performance (e.g. epilepsy, multiple sclerosis, fetal alcohol syndrome).
* Anyone deemed unsafe to study personnel for any reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Marijuana induced performance changes on fMRI Multi-Stage Decision Making (MSDM) Task. | Baseline and post drug administration at 10 minutes.
  The MSDM is a reinforcement learning paradigm that quantifies the degree to which subjects can integrate recent trial-to-trial information about a stimulus' likelihood of reward with acquired knowledge about whether some choices generally lead to disadvantageous outcomes vs. others that more often lead to reward.
Marijuana induced performance changes on Relational and Item Specific Coding (RISE) fMRI Task. | Baseline and post drug administration at 10 minutes.
  The RISE task is a hippocampal-dependent learning paradigm that assesses declarative memory.
Marijuana induced performance changes on fMRI Treadway/Effort Reward Task. | Baseline and post drug administration at 10 minutes.
  The Treadway Effort/Reward Task independently measures the neural responses to two dimensions of a cost/benefit decision: the effort required and the magnitude of reward.
Marijuana induced performance changes on fMRI Monetary Incentive Delay (MID) Task. | Baseline and post drug administration at 10 minutes.
  The MID task probes the brain's reward system to assess the anticipation and receipt of rewards or punishment.

CONTACTS AND LOCATIONS:
Overall Officials: Godfrey Pearlson, M.D, Principal Investigator — Yale University
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States